CLINICAL TRIAL: NCT02022267
Title: Results of Gait Analysis Including Oxford Foot Model in Children With Clubfoot Treated With the Ponseti Method
Brief Title: Gait Analysis in Ponseti Clubfoot
Status: Completed | Type: Observational
Sponsor: Orthopedic Hospital Vienna Speising (Other)
Responsible Party: Principal Investigator, Christof Radler, Assoc. Prof., MD, Orthopedic Hospital Vienna Speising
Other Study IDs: EK10-218-1210
Record Dates: First submitted 2013-12-07; First posted 2013-12-27 (Estimated); Last update posted 2013-12-27 (Estimated); Status verified 2013-12

CONDITIONS: Clubfoot
Keywords: clubfoot; gait analysis; outcome questionaire; Ponseti method
MeSH Terms: conditions — Clubfoot

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- study group: Patients with a minimum age of three years from our prospective, consecutive database of patients with clubfoot treated with the Ponseti method beginning in 2002 are considered for this study. Patients with unilateral or bilateral idiopathic clubfoot are included. Patients with clubfoot associated with syndromes or neurological diseases, with mild clubfoot that required fewer than three casts for initial correction, who first presented at an age older than three months, who were living outside of the country, and who were initially treated elsewhere with more than three casts are excluded.
- control group: healthy children of employees of our hospital

SUMMARY:
Patients with clubfoot treated with the Ponseti method from a prospective database are evaluated using gait analysis including a foot model and a disease specific instrument score and compared to a group of healthy children.

DETAILED DESCRIPTION:
Patients with a minimum age of three years from a prospective, consecutive database of patients with clubfoot treated with the Ponseti method beginning in 2002 are considered for this study. Thereby patients will typically have a follow up of nearly three to eight years after initial clubfoot correction. Patients with unilateral or bilateral idiopathic clubfoot are included. Patients with clubfoot associated with syndromes or neurological diseases, with mild clubfoot that required fewer than three casts for initial correction, who first presented at an age older than three months, who were living outside of the country, and who were initially treated elsewhere with more than three casts are excluded. An invitation letter to participate in the study was sent out at the end of 2011, with a second letter being sent out three months after the first. After the second letter patients had a time frame of three more months to participate before the study was closed.

To comprise a control group for the purpose of collecting gait analysis data of healthy children, employees of our hospital are asked to allow their children to participate in this study.

Each patient will be physically examined, active and passive range of motion (ROM) of the ankle joint will be measured with a hand-held goniometer. Ability to walk on the heels and on tiptoes will be recorded. The disease-specific instrument questionnaire, which will be blinded for the treating physician will be handed out to fill in.

Patients will undergo gait analysis, including video recordings with a Vicon motion capture system (Vicon, Oxford, UK) with kinetic data collected from three AMTI force plates (Advanced Mechanical Technology, Inc., Watertown, MA). Placement of markers will be a combination of Cleveland (lower extremity), PlugInGait (upper body), and Oxford Foot (movement within the foot) models.

ELIGIBILITY:
Inclusion Criteria:

* unilateral or bilateral idiopathic clubfoot treated with the Ponseti method

Exclusion Criteria:

* clubfoot associated with syndromes or neurological diseases
* mild clubfoot that required fewer than three casts for initial correction
* clubfoot patients that first presented at an age older than three months
* clubfoot patients who were living outside of the Country
* clubfoot patients who were treated elsewhere with more than three casts

Ages: 3 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Patients with a minimum age of three years from a prospective, consecutive database of patients with clubfoot treated with the Ponseti method beginning in 2002
Sampling Method: Non-Probability Sample
Enrollment: 51 (Actual)
Dates: Start 2011-10; Primary Completion 2012-02 (Actual); Study Completion 2012-09 (Actual)

PRIMARY OUTCOMES:
3D Gait Analysis with foot model | once at time of presentation for study specific examination; invitations were sent out end of 2011, a second letter three months after the first. After second letter patients had a time frame of three more months to participate before study was closed
  Gait analysis, including video recordings with a Vicon motion capture system (Vicon, Oxford, UK) with kinetic data collected from three AMTI force plates (Advanced Mechanical Technology, Inc., Watertown, MA). Placement of markers will be a combination of Cleveland (lower extremity), PlugInGait (upper body), and Oxford Foot (movement within the foot) models.

SECONDARY OUTCOMES:
Clinical examination | once at time of presentation for study specific examination; invitations were sent out end of 2011, a second letter three months after the first. After second letter patients had a time frame of three more months to participate before study was closed
  Active and passive range of motion (ROM) of the ankle joint measured with a hand-held goniometer. Ability to walk on the heels and on tiptoes.
disease-specific instrument questionnaire | once at time of presentation for study specific examination; invitations were sent out end of 2011, a second letter three months after the first. After second letter patients had a time frame of three more months to participate before study was closed
  questionnaire as described in citation

CONTACTS AND LOCATIONS:
Overall Officials: Christof Radler, MD, Principal Investigator — Orthopaedic Hospital Speising
Locations (1):
- Orthopaedic Hospital Speising, Vienna, Austria

REFERENCES:
- [Background] Roye BD, Vitale MG, Gelijns AC, Roye DP Jr. Patient-based outcomes after clubfoot surgery. J Pediatr Orthop. 2001 Jan-Feb;21(1):42-9. doi: 10.1097/00004694-200101000-00010. PMID 11176352